CLINICAL TRIAL: NCT02984423
Title: Frontline Approach for BRCA Testing in OC Treatment naïve Population. A LATIN AMERICA Epidemiologic Study
Brief Title: FLABRA: Frontline Approach for BRCA Testing in OC Treatment naïve Population. A LATIN AMERICA Epidemiologic Study
Acronym: FLABRA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0817R00002
Record Dates: First submitted 2016-11-23; First posted 2016-12-07 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; BRCA mutations
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archived tumor blocks or twenty 10-µm sections from eligible patients will be requested from the local pathology lab and used for BRCA mutations testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to answer very important questions regarding the prevalence of somatic and germline mutations (sBRCAm and gBRCAm) in a population of newly diagnosed ovarian cancer patients from Latin America. These answers may be extremely helpful in the counseling for genetic risk and treatment approach in these populations and will aid in making treatment decisions in the future

DETAILED DESCRIPTION:
FLABRA is a cross-sectional, multi-center, epidemiological observational study designed to evaluate the prevalence of BRCA mutations in newly diagnosed ovarian cancer patients across understudied ethnic groups in Latin America. Secondary objectives of the study are to evaluate the prevalence of sBRCAm versus gBRCAm in newly diagnosed ovarian cancer patients and to describe current ovarian cancer counselling and treatment approach patterns at front line setting across Latin America.

In the Screening Visit, consecutive eligible patients who have been newly diagnosed with ovarian cancer within the last 120 days will be invited to participate. After having provided consent, patients will be asked to provide ethnicity and cancer family history information. Patients will self-identify to one or more of the defined broad ethnic groups (Native American, Afro-Caribbean, Caucasian) based on self-reported ancestry information. Archived tumor blocks or twenty 10-µm sections from eligible patients will be requested from the local pathology lab and used for BRCA mutations testing.

Patient medical records will be reviewed for data relevant to the ovarian cancer diagnosis, including basic demographics, medical history, and treatment history.

During the Devolution Visit, results of the tumor BRCA test will be communicated to the patient, and information about counselling approach and treatment plan will be recorded in the medical chart. This Devolution Visit will be the last visit for this study for the cases of non-mutated patients. For patients for whom a BRCA mutation have been identified in tumor, additional test in blood looking for the specific point mutation found in tumor will be performed to investigate if these patients harbor a germline BRCA mutation. For these patients a further visit will be organised to communicate results to the patient and data regarding germline test results will be recorded in the medical chart of the patient.

ELIGIBILITY:
Inclussion criteria:

1. Be able and willing to sign the informed consent form
2. Be older than 18 years of age
3. Have histologically confirmed new diagnosis of Federation of Gynecology and Obstetrics stage III or IV ovarian epithelial, primary peritoneal, or fallopian tube cancer made by one or more of the following:

   * standard staging laparotomy including bilateral salpingo-oophorectomy, omentectomy, and lymph node sampling and debulking and or
   * surgical resection and radiographic evidence consistent with Stage 3 or 4 ovarian cancer
   * paracentesis or biopsy with radiographic evidence consistent with Stage III or IV ovarian cancer (normal appearing pancreas, liver, and gastrointestinal tract)
4. Have availability of paraffin-embedded archived tumor tissue block (preferred) or, if a block is not possible, a minimum of twenty 10 microm sections
5. Have a diagnosis that is within 120 days of informed consent

Exclusion criteria:

1. Have a diagnosis of any severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of the study results and, in the judgement of the Investigator, would make the patient inappropriate for enrollment in this study
2. Be a patient who, in the judgement of the Investigator, would be inappropriate for enrollment in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed patients with (FIGO) stage III or IV ovarian epithelial, primary peritoneal, or fallopian tube cancer made
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of BRCA 1 and BRCA 2 mutations in newly diagnosed ovarian cancer patients from Latinoamerican population | up to one year
  FLABRA is a cross-sectional, multi-center, epidemiological observational study designed to evaluate the prevalence of BRCA mutations in newly diagnosed ovarian cancer patients across understudied ethnic groups in Latin America

SECONDARY OUTCOMES:
Prevalence of somatic and germline BRCA 1 and 2 mutations across Latinamerican population | up to one year
  To estimate the prevalence of gBRCAm in newly diagnosed ovarian cancer patients who have a BRCA mutation identified in the tumor sample, in LATAM population, and by ethnic sub-groups
Counselling approach in ovarian cancer across Latinamerican countries | up to one year
  To describe all professionals participating in this process, and time for the approach

CONTACTS AND LOCATIONS:
Locations (22):
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, La Rioja
  - Research Site, Resistencia
  - Research Site, Rosario
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Jaú
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Colombia (3):
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Medellín
- Research Site, México, Mexico
- Research Site, Panama City, Panama
- Peru (2):
  - Research Site, Lima
  - Research Site, San Isidro

REFERENCES:
- [Derived] Giornelli G, Gallardo D, Hegg R, Abuin GG, La Vega M, Lim-Law M, Caceres V, Trujillo L, Pilar Estevez-Diz MD, Pacheco C, Sganga L, Goncalves S. FLABRA, frontline approach for BRCA testing in an ovarian cancer population: a Latin America epidemiologic study. Future Oncol. 2021 May;17(13):1601-1609. doi: 10.2217/fon-2020-1152. Epub 2021 Jan 8. PMID 33415992
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0817R00002&attachmentIdentifier=34f1602d-4fbf-424b-b632-55352d326864&fileName=20200708_FLABRA_CSR_summary.pdf&versionIdentifier=